CLINICAL TRIAL: NCT06546280
Title: Camrelizumab Plus Apatinib as Adjuvant Therapy in Patients With Hepatocellular Carcinoma at High Risk of Recurrence After Radical Resection or Ablation: a Single-arm, Single-center, Exploratory Trial
Brief Title: A Study of Camrelizumab Plus Apatinib as Adjuvant Therapy in Patients With Hepatocellular Carcinoma at High Risk of Recurrence After Radical Resection or Ablation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-220-01
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: Camrelizumab; Drug: Apatinib

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200 mg will be administered by IV infusion on Day 1 of each 21-day cycle.
Drug: Apatinib — Apatinib 250 mg will be taken orally once daily.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of camrelizumab plus apatinib as adjuvant therapy for patients with hepatocellular carcinoma at high risk of recurrence after radical resection or ablation.

DETAILED DESCRIPTION:
Postoperative adjuvant therapy is an important means to effectively reduce the risk of hepatocellular carcinoma recurrence and improve survival, but at this stage, there is no globally recognized postoperative adjuvant therapy for HCC. As a new first-line therapeutic agent for advanced hepatocellular carcinoma, camrelizumab plus apatinib has shown good anti-tumor efficacy in the treatment of advanced hepatocellular carcinoma in the CARES-310 study. Therefore, we wanted to explore the efficacy and safety of camrelizumab plus apatinib in adjuvant therapy for patients with hepatocellular carcinoma at high risk of recurrence after radical resection or ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily join this study and sign informed consent form;
* Age≥18 years, male or female;
* Patients were diagnosed with hepatocellular carcinoma by histology or pathology or clinical diagnostic criteria for hepatocellular carcinoma in the "Guidelines for the Diagnosis and Treatment of Primary Liver Cancer (2024 Edition)", and have undergone radical resection or ablation for hepatocellular carcinoma;
* No macrovascular invasion (allowing intraoperative or postoperative pathologic findings of Vp1/Vp2 type portal vein invasion) or extrahepatic metastases assessed by imaging prior to radical treatment;
* Have high-risk recurrence risk factors, the assessment of which should be based on pre-procedure/ablation imaging;
* Child-Pugh liver function classification: Grade A;
* ECOG PS score: 0-1;
* Full recovery from surgical resection or ablation within 4 weeks prior to enrollment.
* Have not received anti-tumor treatment for hepatocellular carcinoma before enrollment, including systemic treatment and local treatment (except for 1-2 times of prophylactic TACE or HAIC treatment 4-8 weeks after radical treatment);
* Patients who underwent radical therapy are allowed to receive 1-2 prophylactic TACE/HAIC treatments (as needed, not mandatory) 4-8 weeks postoperatively, and are required to have fully recovered from TACE/HAIC within 4 weeks prior to receiving study treatment;
* Patients infected with hepatitis B virus (HBV) who started anti-HBV treatment at the screening stage and are willing to receive antiviral treatment (according to local guidelines, e.g., entecavir, etc.) throughout the study period and be monitored regularly can be included; Hepatitis C virus (HCV) ribonucleic acid (RNA)-positive patients must receive antiviral treatment according to guidelines and have a liver function within the CTCAE grade 1 elevation;
* For female patients of childbearing potential and male patients whose partners are women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use reliable and effective contraceptive methods for at least 120 days from the time of signing the informed consent form until the last dose of study drug.
* Adequate hematologic and organ function.

Exclusion Criteria:

* Known sarcomatoid hepatocellular carcinoma, mixed hepatocellular carcinoma and cholangiocarcinoma or fibrolamellar hepatocellular carcinoma;
* History of other malignant tumors within 5 years or simultaneously;
* Severe functional impairment of other vital organs such as heart, brain, lung and kidney;
* Immune deficiency or active autoimmune disease or history of autoimmune disease and the disease may relapse;
* Evidence of tumor recurrence or metastasis before enrollment;
* History of hepatic encephalopathy;
* Known hypersensitivity to the active ingredients and excipients contained in the investigational drugs (camrelizumab, apatinib) of this study, or known history of severe allergy to any other monoclonal antibody or anti-angiogenesis targeted drug;
* Patients with active or history of interstitial pneumonitis or interstitial lung disease requiring hormonal therapy, or pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), pneumoconiosis, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan that may interfere with the detection and management of immune-related pulmonary toxicity; patients with severely impaired lung function; previous radiation pneumonitis in the radiation field is allowed; patients with active tuberculosis;
* Cardiac clinical symptom or cardiovascular disease that is not well controlled;
* History of gastrointestinal hemorrhage or clear tendency of gastrointestinal haemorrhage within 6 months prior to the start of study treatment;
* Severe infection within 4 weeks prior to the start of study treatment; therapeutic antibiotics given orally or intravenously within 2 weeks prior to the start of study treatment;
* Immunosuppressive or systemic hormone therapy for immunosuppression (dose >10 mg/day prednisone or other equipotent hormone) within 14 days prior to the start of study treatment;
* Patients who are preparing for or have previously received an organ or allogeneic bone marrow transplantation;
* Subjects with hypertension that is not well controlled or history of hypertensive crisis or hypertensive encephalopathy;
* Significant vascular disease (eg, aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to the start of study treatment; ular heparin is permitted)
* Known genetic or acquired hemorrhage (e.g., coagulation disorders) or thrombotic tendency, such as hemophiliacs; current or recent (within 10 days prior to start of study treatment) use of full-dose oral or injectable anticoagulant or thrombolytic medications for therapeutic purposes (prophylactic use of low-dose aspirin, low-molecular heparin is permitted)
* Abdominal fistula, gastrointestinal perforation, or abdominal abscess within 6 months prior to the start of study treatment;
* History of intestinal obstruction and or history of clinical signs or symptoms of gastrointestinal obstruction;
* Thrombosis or thromboembolic event within 6 months prior to the start of study treatment, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism, etc.
* Treatment with a live attenuated vaccine within 28 days prior to the start of study treatment or anticipation of need for such a vaccine during treatment with camrelizumab or within 60 days of the final dose of camrelizumab;
* Pregnant or breastfeeding patients;
* Patients who, in the judgment of the investigator, have other factors that may affect the results of the study or cause forced termination of this study, such as alcoholism, drug abuse, other serious illnesses (including psychiatric illnesses) that require comorbid treatment, and serious laboratory abnormalities accompanied by familial or social factors, which would affect the safety of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-08-26 (Estimated); Primary Completion 2026-08-26 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence free survival rate | Assessed up to 12 months
  Proportion of patients who did not experience recurrence of hepatocellular carcinoma within 1 year of enrollment

SECONDARY OUTCOMES:
Recurrence free survival | Assessed up to 24 months
  Time from enrollment to first occurrence of intrahepatic or extrahepatic hepatocellular carcinoma or death from any cause
Time to recurrence | Assessed up to 24 months
  Time from enrollment to first occurrence of intrahepatic or extrahepatic hepatocellular carcinoma
Overall survival | Assessed up to 24 months
  Time from enrollment to death of any cause
2-year recurrence free survival rate | Assessed up to 24 months
  Proportion of patients with no recurrence of hepatocellular carcinoma within 2 years of enrollment
Adverse events | Assessed up to 12 months
  Includes type, incidence, severity, onset and end time, correlation with treatment/drugs, and regression; severity was graded according to NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Mingxin Pan, Principal Investigator — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No